CLINICAL TRIAL: NCT04115930
Title: Correlation Between Daily Physical Activity and Disability, Fatigue, Cognition and Quality of Life in MS Patients
Acronym: PAMS
Status: Completed | Type: Observational
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Other Study IDs: PAMS
Record Dates: First submitted 2019-04-04; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Fatigue; Quality of Life; Physical Activity
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Fatigue, cognition and quality of life measurements with different kind of tests and forms. EDSS and SFMC. Daily physical activity measurement 7days. Berg´s scale. Sit-Up 30 s and 6-minutes walking test. Length, weight and waist measurements.
  Interventions: Device: Physical Activity measurement:
- Control: Healthy volunteers. Fatigue, cognition and quality of life measurements with different kind of tests and forms. SFMC. Daily physical activity measurement 7days. Berg´s scale. Sit-Up 30 s and 6-minutes walking test. Length, weight and waist measurements.
  Interventions: Device: Physical Activity measurement:

INTERVENTIONS:
Device: Physical Activity measurement: — 7 days measurement with Active style Pro HJA-350IT device

SUMMARY:
The main purpose of the study is to assess the fatigue, cognition, quality of life and disability correlation to MS-patients daily physical activity.

ELIGIBILITY:
Inclusion Criteria:

* RR-MS (relapsing-remitting MS-disease)
* Age 18-55y
* Expanded Disability Status Scale (EDSS) score less than equals to (<=) 5.5
* Not relapse in previous month
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* PP-MS (primary progressive disease)
* SPMS (secondary progressive disease)
* Other protocol defined exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient group: RRMS patients (18-55 years old)
  Control group: Healthy volunteers (18-55 years old)
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Correlation between daily physical activity and quality of life to disability. | Baseline (one measurement)
  Daily physical activity will be measured 7 days assessed by ActiGraphTM wGT3X-BT. Person keep this on his/her wake-up time whole 7 days excluding time when she/he is in water like in shower or swimming. Quality of life will be assessed by questionnaires 15-D and RAND-36 and disability will be assessed by EDSS (Expanded Disability Status Scale) and also with MSFC (Multiple Sclerosis Functional Composite) measurement.
Correlation between fatigue and cognition to daily physical activity and disability. | Baseline (one measurement)
  Fatigue will be assessed with two different questionnaires FSS (fatigue severity scale) and MFIS (Modified Fatigue Impact Scale). Cognition will be assessed SDMT (Symbol Digital Modality Test) and PASAT-test. Daily physical activity will be measured 7 days with measure ActiGraphTM wGT3X-BT. Person keep this on his/her wake-up time whole 7 days excluding time when she/he is in water like in shower or swimming. Disability will be assessed EDSS (Expanded Disability Status Scale) and also with MSFC (Multiple Sclerosis Functional Composite) measurement.
Correlation between fatigue, cognition, quality of life and daily physical activity. | Baseline (one measurement)
  Fatigue will be assessed with two different questionnaires FSS (fatigue severity scale) and MFIS (Modified Fatigue Impact Scale). Cognition will be assessed SDMT (Symbol Digital Modality Test) and PASAT-test. Quality of life will be assessed questionnaires 15-D and RAND-36. Daily physical activity will be measured 7 days with measure ActiGraphTM wGT3X-BT. Person keep this on his/her wake-up time whole 7 days excluding time when she/he is in water like in shower or swimming.
Disability level EDSS | Baseline (one measurement)
  Disability will be assessed EDSS (Expanded Disability Status Scale). Scale range is between 0 to 10. (0 level is normal and 10 means death)
Disability level MSFC | Baseline (one measurement)
  Disability will be assessed MSFC (Multiple Sclerosis Functional Composite) measurement. Test include three different kind of test The Timed 25-Foot Walk Test, The 9-HPT (9-hole peg test) and The Paced Auditory Serial Addition Test "PASAT"). The MSFC is based on the concept that scores for these three dimensions-arm, leg, and cognitive function are combined to create a single score (the MSFC) that can be used to detect change over time in a group of multiple sclerosis patients. This is done by creating Z-scores for each component of the MSFC and averaging them to create an overall composite score known as the MSFC score. ex. MSFC Score = {Zarm, average + Zleg, average + Zcognitive} / 3.0 Where Zxxx =Z-score
9-Hole Peg Test | Baseline (one measurement)
  The 9-HPT (9-hole peg test). The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and non-dominant hands are tested twice (two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand). Record only the times for the two successfully completed trials for each hand. (time/within 0.1 seconds,lower time is better.)
The Timed 25-Foot Walk test | Baseline (one measurement)
  The Timed 25-Foot Walk test is a quantitative measure of lower extremity function. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible. Record the subject's walk time to within 0.1 second, lower time is better)
Daily physical activity | 7 days
  Daily physical activity will be measured 7 days with measure ActiGraphTM wGT3X-BT. Person keep this on his/her wake-up time whole 7 days excluding time when she/he is in water like in shower or swimming.
Quality of life 15-D | Baseline (one measurement)
  Quality of life level will be assessed questionnaire 15-D. 15 question (evaluation 5 class in every question= 1 to 5 points) Count together and higher number is worse.
Quality of life RAND-36 | Baseline (one measurement)
  Quality of life level will be assessed questionnaire RAND-36.(include 36 question in 8 different kind of section). Higher number is worse.
Cognition level SDMT | Baseline (one measurement)
  Cognition will be assessed with SDMT (Symbol Digital Modality Test). Higher number is better.
Cognition level PASAT | Baseline (one measurement)
  Cognition will be assessed with PASAT-test.(Paced Auditory Serial Addition Test). The test score is the number of correct sums given (out of 60 possible) in each trial. Higher number is better.
Fatigue level FSS | Baseline (one measurement)
  Fatigue will be assessed with questionnaire FSS (fatigue severity scale). FSS questionaire containing nine statements that attempt to explore severity of fatigue symptoms. The subject is asked to read each statement and circle a number from 1 to 7. The scoring is done by calculating the average response to the questions (adding up all the answers and dividing by nine). Higher number is worse.
Fatigue level MFIS | Baseline (one measurement)
  Fatigue will be assessed with questionnaire MFIS (Modified Fatigue Impact Scale). 21 questions. (scale 0 to 4 in every questions/ range 0 to 84 in whole questionnaire). Higher number is worse.
General condition (endurance) | Baseline (one measurement)
  General condition (endurance) assessed by 6-minutes walking test distance in meters.

SECONDARY OUTCOMES:
Body Composition Weight | Baseline (one measurement)
  Body composition evaluation assesment by weight (kg)
Body Composition Height | Baseline (one measurement)
  Body composition evaluation assesment by height (cm)
Body Composition Weist | Baseline (one measurement)
  Body composition evaluation assesment by weist (cm)
Body Composition BMI | Baseline (one measurement)
  BMI (Body Mass index). Weight and height will be combined to report BMI in kg/m^2
Equilibrioception (balance) | Baseline (one measurement)
  Equilibrioception evaluation by Berg´s balance scale. 14 different part and scale in every part 0 to 4. Count together and whole test range 0 to 56. (Higher is better)
Abs strength | Baseline (one measurement)
  Abs strength assessed by 30 seconds sit-ups (amount)

CONTACTS AND LOCATIONS:
Overall Officials: Marko Luostarinen, Principal Investigator — University of Eastern Finland
Locations (4):
- Finland (4):
  - Joensuu, Joensuu
  - Jyväskylä, Jyväskylä
  - University of Eastern Finland, Kuopio
  - Oulu, Oulu

REFERENCES:
- [Derived] Luostarinen M, Portaankorva AM, Urpilainen P, Takala S, Venojarvi M. Correlation of Cognition With Disability and Physical Performance in Patients With Relapsing-Remitting MS. J Cent Nerv Syst Dis. 2025 Jun 17;17:11795735251349716. doi: 10.1177/11795735251349716. eCollection 2025. PMID 40535778